CLINICAL TRIAL: NCT04591184
Title: Phase I/II Study to Evaluate Safety, Tolerability, and Immunogenicity of a Prophylactic Plasmid DNA Vaccine Against SARS-CoV-2 [Covigenix VAX-001/VAX-001-1b] in Healthy Adults 18 Years and Older
Brief Title: A Clinical Trial of a Prophylactic Plasmid DNA Vaccine for COVID-19 [Covigenix VAX-001] in Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Entos Pharmaceuticals Inc. (Industry)
Collaborators: Aegis Life, Inc. (Unknown); Canadian Institutes of Health Research (CIHR) (Other Government); Clinical Pharma Solutions Inc (Unknown); Centre national de recherche et de formation sur le paludisme (CNRFP) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ENTVAX01-101
Record Dates: First submitted 2020-09-23; First posted 2020-10-19 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: SARS-CoV-2
Keywords: COVID-19; SARS-CoV-2; anti-infective; prophylaxis; healthy volunteer; prevention; Covigenix VAX-001
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Unblinded study nurse with no other role in the trial administers VAX-001. Observer blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Covigenix VAX-001 (Experimental): Dose-ranging, 2 dose levels. 24 subjects receiving active i.m. vaccine
  Interventions: Biological: Covigenix VAX-001
- Placebo (Placebo Comparator): Placebo injection. 12 subjects receiving placebo
  Interventions: Biological: Covigenix VAX-001 placebo

INTERVENTIONS:
Biological: Covigenix VAX-001 placebo — Placebo vaccine
  Arms: Placebo
Biological: Covigenix VAX-001 — Active Covigenix VAX-001
  Arms: Active Covigenix VAX-001

SUMMARY:
This study is a Phase I/II clinical study in healthy adults designed to assess the safety, tolerability, and immunogenicity of receiving 2 IM injections of Covigenix VAX-001/-1b, 28 days apart. Covigenix VAX-001/-1b is a plasmid DNA vaccine that expresses key antigenic determinants from SARS-CoV-2 and uses Entos Pharmaceuticals' Fusogenix PLV platform.

The phase I part of this study was completed in Canada. The phase II part of the study will be completed in Burkina Faso, Senegal and South Africa.

DETAILED DESCRIPTION:
Phase I portion of the study:

Study design:

ENTVAX01-101 is a phase I/II, placebo-controlled, randomized, observer-blind, dose ranging clinical trial in males and non-pregnant females, 18 years and older, who are in good health and meet all eligibility criteria. This clinical trial is designed to assess the safety, tolerability, and immunogenicity of Covigenix VAX-001 manufactured by Entos Pharmaceuticals. Covigenix VAX-001 is a novel plasmid DNA-based vaccine that encodes for the full-length Spike protein from SARS-CoV-2 (VAX-001 encapsulated in a proprietary Fusogenix Proteo-Lipid Vehicle (PLV)).

Enrollment for the phase I portion of the study will occur at one Canadian site. Thirty-six participants will be enrolled in a staggered manner into one cohort an 3 groups (0.100 mg & 0.250 mg vs. placebo) in stage I. Participants will receive an intramuscular (IM) injection (0.5 milliliter [mL]) on Days 0 and 14 in the deltoid muscle of alternating arms and will be followed through 12 months post booster vaccination (Day 379). Follow-up visits will occur at Days 7, 14, 17, 21, 28, 42, 196, and 379.

The primary objective is to evaluate the safety of a 2-dose vaccination schedule of the Covigenix VAX-001 vaccine, given 14 days apart. The secondary objectives are to evaluate the humoral immune response as measured by Immunoglobulin G (IgG) ELISA to the SARS-CoV-2 S protein and by pseudo-viral neutralization assay to pseudo-virion following a 2-dose vaccination schedule of Covigenix VAX-001.

Clinical safety data will be collected at the Day 0 of the study and at defined intervals (Dose 1: Days 7, 14; Dose 2: Days: 21, 42).

Clinical safety lab testing

• Hematology & Biochemistry:

Immunogenicity testing:

* ELISA and pseudo-viral neutralization tests
* % of responders or individuals who seroconvert (with 95% CI): develop immune response defined as a 4-fold or greater rise.
* Geometric mean concentration/geometric mean titers (with 95% CI) and pre-/post-vaccination ratios (geometric mean ratios) provide absolute values and increase in antibody titers at defined time points after each vaccination.
* Reverse cumulative distribution (RCD) curves display percentage of participants versus antibody levels.

The following immunogenicity tests will be performed as exploratory objectives:

* SARS-CoV-2 neutralization antibody responses at Days 0, 7, 14, 21, 28, 42, 196, and 379.
* Antigen-specific B&T cell interferon (IFN)-γ cell responses measured by ELISPOT up to Day 379.
* Antigen-specific T cell responses measured by flow cytometry up to Day 379
* Antigen-specific T cell responses including cluster of differentiation (CD)4+ and CD8+ cytotoxic T lymphocytes (CTLs), through ICS up to Day 379
* Whole blood immunophenotyping (B and T cell repertoire (BCR and TCR) as measured by high throughput sequencing of lymphocyte antigen receptor genes, SCS, and RNAseq to identify all genes regulated by the vaccine) up to Day 379

Sample size: 36 participants, 24 test subjects and 12 placebo controls;

Study plan:

Table 1. Study groups and treatments Arm Intervention

1. Experimental: Low dose (0.100mg), 18-<55 years, 2 doses Biological: Covigenix VAX-001, 0.5 mL IM injection
2. Experimental: High dose (0.250mg), 18-<55 years, 2 doses Biological: Covigenix VAX-001, 0.5 mL IM injection
3. Placebo Comparator: Placebo, 18-<55 years Other: Placebo, 0.5 mL IM injection

Enrollment plan:

Enrollment plan: Study participants will be enrolled in a staged manner at each dosage level (Low and High), as described below:

First, three participants of the cohort will be randomized (2:1; Groups 1 and 3) to the low dose of Covigenix VAX-001 or placebo, a minimum of one hour apart. Once three participants have received treatment there will be a 72-hour waiting period, and if no holding rule is met then the remaining participants from Group 1 and 3 will be vaccinated. Similarly, once 7-day safety data are available on a minimum of 75% (n=14) of participants in Groups 1/3, 1) participants of the cohort will be randomized (2:1; groups 2 and 3) to the high dose of Covigenix VAX-001 or placebo.

After review of day 42 data (Day 28 post second dose) on participants in Groups 1/3 (Low dose), it will be decided whether this group will be enrolled in the Ph II of the study.

Infection during the study: During the observation period of the study, if fever and respiratory symptoms with cough develop in a participant, he/she should immediately follow local procedures for care of suspected COVID-19 illness and contact the study team. The participant's nasopharyngeal and throat swab/sputum will be collected and tested for SARS-CoV-2 at a designated provincial testing center. If a COVID-19 infection is found during the study, a case investigation will be undertaken. Careful monitoring for vaccine-related enhanced disease will be undertaken in conjunction with the participant's primary physician.

In addition to the real-time PCR testing for SARS-CoV-2, the collected nasopharyngeal swab/sputum will be tested for other respiratory pathogens.

Participants testing positive for SARS CoV 2 between IP Dose 1 and Dose 2 will not receive Dose 2, but will be followed for safety.

Study duration: 13 months

Study Design for the phase II portion of the study:

For the Phase II part, enrollment will occur at sites globally. Approximately 500 participants will be enrolled into 1 of 5 groups (approximately 100 per group) as safety data emerge from the Phase I portion . Participants will receive an IM injection (0.5 mL) on Days 0 and 14 in the deltoid muscle of alternating arms and will be followed through 12 months post Dose 2. Follow-up visits will occur at Days 14, 28, 42, 196, and 379.

The total duration for an individual participant in the Phase II part will be approximately 13 months.

Study arms are:

1. Experimental: Low dose (0.100mg), 18 years and older, 2 doses active Biological: Covigenix VAX-001, 0.5 mL IM injection
2. Experimental: Low dose (0.100mg), 18 years and older, 1 dose active, 1 dose placebo Biological: Covigenix VAX-001, 0.5 mL IM injection
3. Experimental: High dose (0.250mg), 18 years and older, 2 doses active Biological: Covigenix VAX-001, 0.5 mL IM injection
4. Experimental: High dose (0.250mg), 18 years and older, 1 dose active, 1 dose placebo Biological: Covigenix VAX-001, 0.5 mL IM injection
5. Placebo Comparator: Placebo, 18 years and older Other: Placebo, 0.5 mL IM injection

Clinical safety lab testing

• Hematology & Biochemistry:

Immunogenicity testing:

* ELISA and pseudo-viral neutralization tests
* % of responders or individuals who seroconvert (with 95% CI): develop immune response defined as a 4-fold or greater rise.
* Geometric mean concentration/geometric mean titers (with 95% CI) and pre-/post-vaccination ratios (geometric mean ratios) provide absolute values and increase in antibody titers at defined time points after each vaccination.

The following immunogenicity tests will be performed as exploratory objectives:

* SARS-CoV-2 neutralization antibody responses at Days 0,14, and 28.
* Antigen-specific T cell responses including cluster of differentiation (CD)4+ and CD8+ cytotoxic T lymphocytes (CTLs), through ICS up to Day 379

Phase II

The Phase II part will be initiated following DSMC recommendation based on 42-day reviews of each group (complete or partial group) in Phase I Canada part and the enrollment and DSMC recommendations from the Phase II Lead-in groups in South Africa, Burkina Faso, and Senegal. Recruitment will be staggered by group as summarized in Table 5 of the protocol. The Phase II part will consist of a randomized, observer-blinded, multi-center, dose ranging clinical study in males and nonpregnant females, 18 years and older who meet all eligibility criteria. Approximately 500 participants will be enrolled into 1 of 4 cohorts: low dose 0.100 mg as 1 or 2 dose schedule and high dose 0.250 mg as 1 or 2 dose schedules.

Participants will receive an IM injection (0.5 mL) on Days 0 and 28 in the deltoid muscle of alternating arms and will be followed through 12 months post Dose 2 (Table 5).

Follow-up visits will occur at Days 28, 42, 56, 118, 210, and 393. Enrollment in the phase II part of the study will be carried out globally in Burkina Faso, Senegal and South Africa.

ELIGIBILITY:
Inclusion Criteria

Inclusion criteria for Phase I:

Each participant must meet all of the following criteria to be enrolled in the Phase 1 part of the study:

1. The participant is a healthy adult from 18 <55 years and with a BMI of ≤30 kg/m2 at the time of enrollment.
2. If the participant is a WOCBP, she must have practiced adequate contraception for 30 days prior to IP Dose 1, have a negative pregnancy test on the day of IP Dose 1, and have agreed to continue adequate contraception until 90 days after IP Dose 2.
3. If the participant is male, he must agree to continue adequate contraception until 90 days after IP Dose 2.
4. The participant is able to provide consent to participate in the study and has signed an ICF.
5. The participant is able and willing to complete all the scheduled study procedures during the whole study period (approximately 13 months).
6. The participant is generally in good health, as determined by a review of medical history and a physical examination within 14 days prior to IP Dose 1.

Inclusion criteria for Phase II

Each participant must meet all of the following criteria to be enrolled in Phase II part of the study:

1. The participant is 18 years and older.
2. If the participant is a WOCBP, she must have a negative pregnancy test on the day of IP Dose 1, and have agreed to adequate contraception until 90 days after IP Dose 2 administration.
3. If the participant is male, he must agree to continue adequate contraception until 90 days after IP Dose 2
4. The participant can provide consent to participate in and having signed an ICF.
5. The participant is able and willing to complete all the scheduled study procedures during the whole study follow-up period (approximately 13 months).

Exclusion Criteria

Exclusion criteria for Phase I

Participants meeting any of the following criteria will be excluded from Phase I of the study:

1. The participant has history of anaphylaxis to any allergen.
2. The participant has history of seizure disorder, encephalopathy or psychosis.
3. The female participant is pregnant (positive urine pregnancy test), lactating, or plans to become pregnant during the 3 months of enrollment.
4. The participant has a positive test result for HIV or hepatitis B and C.
5. The participant has a positive test results of IgG antibodies against SARS CoV 2 from RCT.
6. The participant has a positive test result of real-time quantitative PCR screening of nasopharyngeal swab/sputum for SARS-CoV-2.
7. The participant has a laboratory (hematological and biochemistry) examination that is out of normal range, or greater than a Grade 1 abnormality and clinically significant as assessed by the investigator including test results for: CBC, PT, PTT, ALT, AST, ALP, T Bil, Cr, lipase, and blood glucose;

   - Transient mild laboratory abnormalities may be rescreened once, and the participant will be excluded if the laboratory repeat test is abnormal as per local laboratory normal values and the investigator's assessment.
8. The participant presents with any acute febrile disease (oral temperature ≥38.0°C) or active infectious disease.
9. The participant has a medical history of SARS-CoV-1.
10. The participant has unstable concomitant underlying conditions.

    - Note: Stable condition defined as: The participant is appropriately managed on consistent disease management, for example participants with well controlled hypertension, adult-onset diabetes, Benign Prostate Hypertrophy (BPH) or hypothyroid disease will be eligible for enrollment. The treatment regimen should be stable for at least 3 months prior to entering the study. Once IP treatment has started, must be willing to maintain all aspects of the treatment regimen and forgo any elective changes in medication or management. Emergency changes in medication or management would be captured as an adverse event.
11. The participant has a history of Guillain-Barre Syndrome or degenerative neurological disorders; a history of autoimmune, inflammatory disease or potential immune-mediated medical conditions (PIMMCs), or any condition that may put the participant at increased risk of safety events
12. The participant has serious cardiovascular diseases, such as arrhythmia, conduction block, history of myocardial infarction, severe hypertension not controlled with medication.
13. The participant has a serious chronic disease such as asthma, diabetes, or thyroid disease.
14. The participant has immunodeficiency, asplenia, or functional asplenia.
15. The participant has a platelet disorder or other bleeding disorder that may cause contraindication for IM injection.
16. The participant has chronic obstructive pulmonary disease, current smoker or vaper.
17. The participant has a history or diagnosis of coagulopathies.
18. The participant has received immunosuppressive medication, cytotoxic therapy, or corticosteroids (excluding corticosteroid spray for allergic rhinitis, surface corticosteroid therapy for acute non-complicated dermatitis) in the last 6 months.
19. The participant received the blood products in last 4 months.
20. The participant has received other investigational drugs within 1 month before Day 0, or planned use during the study period.
21. The participant had prior administration of any live attenuated vaccine within 1 month before Day 0.
22. The participant had prior administration of a subunit or inactivated non SARS CoV 2 vaccine within 2 weeks before Day 0.
23. The participant had prior administration of any other vaccine considered (or being considered) to be protective against SARS-CoV-2 any time before Day 0.
24. The participant had prior participation in other studies involving study intervention containing lipid nanoparticles.
25. The participant has any condition that, in the opinion of the investigator, may interfere with the participant's compliance, evaluation of study objectives, or informed consent process (i.e. medical, psychological, social or other conditions).
26. The participant is at high risk of acquiring SARS-CoV-2 infection due to their surroundings, contacts or circumstances. Explicitly exclude healthcare and essential workers/at risk population.

Exclusion criteria for Phase II

Participants meeting any of the following criteria will be excluded from Phase II part of the study:

1. The participant has history of anaphylaxis to any allergen.
2. The female participant is pregnant (positive urine pregnancy test), lactating, or plans to become pregnant during the next 3 months.
3. The participant has any acute febrile disease (oral temperature ≥38.0°C [100.4ºF]) or active infectious disease on the day of IP administration (participants may be re scheduled).
4. The participant has a medical history of SARS-CoV-1.
5. The participant has a history of immunodeficiency, asplenia, or functional asplenia.
6. The participant has received immunosuppressive medication, cytotoxic therapy, inhaled corticosteroids (excluding corticosteroid spray for allergic rhinitis, surface corticosteroid therapy for acute non-complicated dermatitis) in the last 6 months.
7. The participant has received other investigational drugs within 1 month before first dose administration or planned use during the study period.
8. The participant has received any live attenuated vaccine within 1 month before first dose administration or any inactivated vaccine within 2 weeks before first dose administration.
9. The participant has received prior administration of any other vaccine considered (or being considered) to protect against SARS-CoV-2 any time before study onset.
10. The participant has a history of any medical conditions that place them at higher risk for severe illness due to SARS-CoV-2 including but not limited to asthma, chronic kidney disease being treated with dialysis, chronic lung disease, diabetes, hemoglobin disorders, immunocompromised, liver disease, serious heart conditions, or severe obesity.
11. The participant has any condition that in the opinion of the investigators may interfere with the participants' compliance, evaluation of study objectives, or informed consent process (i.e., medical, psychological, social or other conditions).

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 268 (Actual)
Dates: Start 2021-04-07 (Actual); Primary Completion 2023-12-06 (Actual); Study Completion 2023-12-06 (Actual)

PRIMARY OUTCOMES:
Safety of a 2-dose regimen of VAX-001 when doses are given 14 days apart | Day 0 - 42
  Frequency and Grade (mild, moderate, severe, potentially life-threatening; Gr. 1-4, respectively) of solicited injection site and systemic adverse events and unsolicited systemic adverse events
Mean change from baseline in safety laboratory measures | Day 0 - 42
  Adverse hematology /clinical chemistry parameter changes (mild, moderate, severe, or life-threatening; Gr. 1-4, respectively)
Frequency of treatment-emergent Serious Adverse Events (SAE) throughout the study and up to 12 months post-second dose immunization (Day 379). | Day 0 - 379
  Frequency of serious AEs

SECONDARY OUTCOMES:
Percent seroconversion defined as a 4-fold or greater increase in IgG titers after one or two doses as measured by IgG ELISA | Up to Day 379
  Percent seroconversion post second dose as measured by ELISA
Geometric mean neutralizing antibody titers against pseudo-virion after one and two doses | Up to Day 379
  Geometric mean of antibody titers measured by pseudo-viral neutralization assay.
Percent seroconversion defined as a 4-fold or greater increase in IgG titers after one or two doses as measured by pseudo-viral neutralization assay. | up to Day 379
  Seroconversion as measured by pseudo-viral neutralization
Persistence of IgG antibody titers as measured by ELISA and neutralizing antibody titers measured by pseudo-virion neutralization assay, six months after the second vaccine dose | Up to Day 379
  Maintenance of antibody titers up to 12 months post second dose

CONTACTS AND LOCATIONS:
Overall Officials: Joakem Tazanu Fossung, Study Director — Clinical Pharma Solutions
Locations (4):
- National Center for Research and Training on Malaria, Ouagadougou, Burkina Faso
- Canadian Centre for Vaccinology, Dalhousie University, Halifax, Nova Scotia, Canada
- Institute for Health Research, Epidemiological Surveillance and Training (IRESSEF), Dakar, Senegal
- FARMOVS (PTY) Ltd., Bloemfontein, South Africa

IPD SHARING:
Plan to Share IPD: No